CLINICAL TRIAL: NCT03013023
Title: Early Behavioral and Transaction Interventions on Preterm Infants' and Parents' Biopsychosocial Well-being
Brief Title: Effects of Early Behavioral and Transaction Interventions on Preterm Infants' and Parents' Biopsychosocial Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Investigator, National Defense Medical Center, Taiwan, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1-103-05-165
Record Dates: First submitted 2016-12-29; First posted 2017-01-06 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Early Interventions; Preterm Infants; Parent-Child Relations
Keywords: Behavioral and Transaction Interventions; Parents' Biopsychosocial Well-being; Preterm Infants; Sleep; Salivary cortisol
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Routine care (Placebo Comparator): Control group
  Interventions: Behavioral: Routine care
- Behavioral-support interventions (BS) (Active Comparator): NNS, FT, positional support, and oral sucrose feeding will be provided while infants are undergoing painful procedures
  Interventions: Behavioral: BS
- Parent-infant transaction program (PITP) (Active Comparator): The PITP will be a six-session, one-on-one teaching intervention beginning on day 22 after birth, with four sessions at bedside, and two home-visit sessions within the first month after discharge.
  Interventions: Behavioral: PITP
- BS+PITP (Active Comparator): Behavioral-support interventions + Parent-infant transaction program
  Interventions: Behavioral: BS+PITP

INTERVENTIONS:
Behavioral: BS — NNS, FT, positional support, and oral sucrose feeding
  Arms: Behavioral-support interventions (BS)
Behavioral: Routine care — Routine NICU care
  Arms: Routine care
Behavioral: PITP — Parents will learn to regulate infant responses while implementing caregiving activities.
  Arms: Parent-infant transaction program (PITP)
Behavioral: BS+PITP — Parents will learn to regulate infant responses while implementing caregiving activities. Supportive interventions, i.e., NNS, FT, positional support, and oral sucrose feeding, will be provided while infants are undergoing painful procedures.
  Arms: BS+PITP

SUMMARY:
This randomized controlled trial will use a longitudinal repeated-measures design to examine the effects of two interventions, behavioral support interventions and a parent-infant transactional program, on parents' stress, PPD and sleep quality, parent-infant interactions, and their preterm infants' stress (saliva cortisol levels), sleep patterns, emotional regulation, and neurobehavioral developmental outcomes from 7 days to 2 years corrected age.

DETAILED DESCRIPTION:
The proposed study has five specific aims:

1. to develop behavioral-support interventions for preterm infants who receive painful, stressful procedures in the NICU,
2. to develop a parent-infant transactional program (PITP) for parent-infant dyads with preterm infants in the NICU,
3. to determine the short-term effects of the behavioral-support interventions and PITP on infant stress (salivary cortisol levels) and sleep patterns,
4. to determine the short-term effects of the PITP on parental stress, depression, social support, and sleep quality during postpartum, and
5. to determine the long-term effects of the behavioral-support interventions and PITP on parent-infant interactions and infants' long-term emotional regulation and neurobehavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age (GA) > 28 weeks and < 37 weeks
2. Postbirth age >2 days
3. Stable condition (score<20 on the Neonatal Therapeutic Intervention Scoring System [NTISS] for disease severity).
4. Parents are not diagnosed with mental illness or some other illness known to influence/confound the outcome variables
5. Parents are fluent in Chinese
6. Parents do not use drugs
7. Parents agree to participate in this study

Exclusion Criteria:

1. Congenital anomalies
2. Neurologic impairment including convulsion, intraventricular hemorrhage > grade II or periventricular leukomalacia
3. Documented congenital or nosocomial (infection acquired at hospital after birth) sepsis
4. Surgery
5. Severe medical conditions requiring treatments such as cortisol supplementation, sedatives, muscle relaxants, antiepileptic, or analgesic drugs

Ages: 28 Weeks to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Parent stress | 7days to 12 months
  Accessed by Parenting Stress Index-Short form (PSI-SF)
Parent depression | 7days to 12 months
  Accessed by the Edinburgh Postnatal Depression Scale (EPDS)
Parent sleep | 7days to 12 months
  Accessed by Pittsburgh Sleep Quality Index
Parent social support | 7days to 12 months
  Accessed by the Social Support Rating Scale (SSRS)

SECONDARY OUTCOMES:
Parent-infant interaction | 1 month to 6 months
  Assessed by NCASTfeeding scale
Preterm infant's sleep | up to 3 months
  Assessed by Actigraphy
Preterm infant's stress | up to 3 months
  Assessed by Salivary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Jiuan Liaw, Professor, Study Chair — Professor, School of Nursing, National Defense Medical Center, Taipei, Taiwan, ROC.

IPD SHARING:
Plan to Share IPD: No